CLINICAL TRIAL: NCT01395472
Title: Influence of Physical Exercise on Cognitive Functioning of Traumatic Brain Injury Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Patricia Rzezak PhD, Federal University of São Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TBI-1858/09
Record Dates: First submitted 2011-07-13; First posted 2011-07-15 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-04

CONDITIONS: Brain Injuries; Brain Diseases; Central Nervous System Diseases; Craniocerebral Trauma; Trauma, Nervous System
Keywords: TBI; Acute physical exercise; Cognitive functions; Mood
MeSH Terms: conditions — Brain Injuries; Brain Diseases; Central Nervous System Diseases; Craniocerebral Trauma; Trauma, Nervous System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- TBI - Experimental Sample (Experimental): TBI patients will be submitted to two acute physical exercise protocols in a cycloergometer with one weak of interval (until voluntary exhaustion and 30 minutes in ventilatory threshold I)
  Interventions: Behavioral: Acute Physical Exercise
- Healthy Controls (Active Comparator): healthy volunteers will be submitted to two acute physical exercise protocols in a cycloergometer with one weak of interval (until voluntary exhaustion and 30 minutes in ventilatory threshold I)
  Interventions: Behavioral: Acute Physical Exercise
- TBI Controls (Active Comparator): Patients will be submitted to a protocol of stretching for 30 minutes
  Interventions: Behavioral: Stretching protocol

INTERVENTIONS:
Behavioral: Acute Physical Exercise — Patients and healthy volunteers will be submitted to a protocol of progressive maximal exercise until voluntary exhaustion and one weak later to 30 minutes of physical exercise in ventilatory threshold I, both in the same cycloergometer.
  Arms: Healthy Controls; TBI - Experimental Sample
Behavioral: Stretching protocol — TBI patients will be submitted to 30 minutes of stretching exercises composed of 15 exercises that prioritize back, legs and hip.
  Arms: TBI Controls

SUMMARY:
The aim of this study is to determine the effects of an acute session of physical exercise on cognitive functioning and humor of traumatic brain injury patients and to investigate whether different cognitive responses can be achieved with different intensities of exercise (moderate and vigorous).

The investigators hypothesize that while moderate intensity physical exercise may be beneficial to cognitive functioning, vigorous intensity may be detrimental to TBI patients, as physical fatigue may impair alertness and other higher cognitive functions.

DETAILED DESCRIPTION:
It is well known the benefits of physical exercise to cognitive functioning, which have been demonstrated in animal studies and in those with healthy humans or with individuals with some type of pathology. Nevertheless, there are few studies investigating the effects of acute physical exercise on cognitive functions of people with traumatic brain injury, even though they frequently have impairments in several cognitive domains due to their brain damage.

The effect of two intensities of physical exercise (moderate and exhaustive) in attention, processing speed, memory, executive control and decision making will be investigated in patients with TBI. For that matter, their performance will be compared to non-brain injured subjects submitted to the same protocol and to TBI patients submitted to a stretching session.

Each subject will be submitted to a neuropsychological evaluation before and after the physical exercise in order to determine if there is an improvement in cognitive performance post-exercise.

ELIGIBILITY:
Patients with TBI eligible for participation in this research study must meet the following inclusion criteria:

Inclusion Criteria:

* diagnose of moderate to severe TBI
* be at least six-months post-injury
* have a neurologist that allowed to enroll into the study
* be able to take part in a cycloergometer-protocol, attested by the laboratory (CEPE) physician
* brain injury must have occurred in adult life
* provided written informed consent for participation

Exclusion Criteria:

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-10 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological evaluation | 1 Day
  Neuropsychological evaluation will be held immediately before the execution of physical exercise (maximal, 30 minutes in ventilatory threshold I or stretching exercise) and immediately after the conclusion of exercise.

SECONDARY OUTCOMES:
Mood, fatigue and impulsivity questionnaires | 1 day
  Mood, fatigue and impulsivity questionnaires will be held immediately before the execution of physical exercise (maximal, 30 minutes in ventilatory threshold I or stretching exercise) and immediately after the conclusion of exercise

CONTACTS AND LOCATIONS:
Overall Officials: Marco T De Mello, PhD, Study Chair — Centro de Estudos em Psicobiologia e Exercício/AFIP; Patricia Rzezak, PhD, Principal Investigator — Centro de Estudos em Psicobiologia e Exercício/AFIP
Locations (1):
- Centro de Estudos em Psicobiologia e Exercício/AFIP, São Paulo, São Paulo, Brazil